CLINICAL TRIAL: NCT01601106
Title: A Phase I/II, Single-Center, Randomized, Placebo-Controlled Study Evaluating the Therapeutic Efficacy of Intravenously Injected PEG-liposomal Prednisolone Sodium Phosphate (Nanocort®) in Subjects With Severe Inflamed Carotid or Aortic Atherosclerosis Plaques
Brief Title: Silencing Inflammatory Activity by Injecting Nanocort in Patients at Risk for Atherosclerotic Disease
Acronym: SILENCE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL37190.018.11
Record Dates: First submitted 2011-10-13; First posted 2012-05-17 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Atherosclerosis; Inflammation
Keywords: Atherosclerosis, inflammation
MeSH Terms: conditions — Atherosclerosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Liposomal prednisolone (Active Comparator)
  Interventions: Drug: liposomal prednisolone
- Placebo control (Placebo Comparator)
  Interventions: Drug: liposomal prednisolone; Drug: Placebo

INTERVENTIONS:
Drug: liposomal prednisolone — Two weekly dosages with 150 mg.
Drug: Placebo
  Arms: Placebo control

SUMMARY:
Cardiovascular disease(CVD) is the leading cause of morbidity and mortality in developed nations. CVD is primarily caused by atherosclerosis, a systemic disease characterized by lipid deposition in the subendothelial space with a concomitant, low-grade inflammatory reaction.(Fuster, Moreno et al. 2005) To date, most therapeutic interventions aimed at lowering CVD have thus far focused on modulating lipid levels, either lowering LDLc or increasing HDLc levels. Yet, since the introduction of statins 20 years ago, there have been few breakthroughs in the treatment of this disease. A promising strategy to reduce CVD is to directly target inflammation at the level of the vessel wall.(van Leuven, van Wijk et al.; Libby 2002) A potential drawback of anti-inflammatory strategies pertains to the thin line between inhibiting 'inappropriate' inflammation versus inducing immuno-suppression. Therefore, continuous low dosed anti-inflammatory drugs have great potential as novel treatment strategies. In the present project, the investigators propose to inject liposomal glucocorticoids intravenously in patients with an increased risk of atherosclerotic disease aiming to reduce vessel wall inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Population with target to background ratio of 2.2 of the aorta or carotid artery on PET-CT

Exclusion Criteria:

* Current medical history of auto-immune disease/vasculitis, active inflammatory diseases, Recent (<1 month prior to screening) or ongoing serious infection requiring IV antibiotic therapy.
* Recent or current treatment with medications that may have a significant effect on plaque inflammation as measured by plaque TBR, including but not limited to:

  * Steroids for at least 6 weeks prior to baseline measurement and during study (with the exception of inhaled acute use steroids).
  * Biological based medicines (anti-TNF (ex. Infliximab), anti-IL-6 therapy (ex. Tocilizumab) or anti-IL-1 (ex. anakinra)) within 8 weeks before the baseline visit and during the study
  * No other disease modifying antirheumatic drugs (DMRADS) within 6 weeks of baseline and during study (such as cyclosporine, azatioprine, etc.)
* Known systemic disorders such as hepatic, renal, hematologic, and malignant diseases or any clinically significant medical condition that could interfere with the conduct of the study.
* Changes in dose or frequency of doses at least 6 weeks prior to baseline measurement (unstable dosing) in angiotensin-converting enzyme (ACE) inhibitors (ACE-I) or angiotensin-receptor blockers (ARBs), non-statin lipid-modifying therapy, thiazolidinediones, inhaled steroids, or leukotriene modifying agents, nonsteroidal anti-inflammatory drugs (NSAIDS), and cyclo-oxygenase-2 inhibitors (COXIBs)
* Standard contra-indications to MRI, 18FDG PET, and CT based on physicians experience and current practices
* Current medical history of poorly controlled diabetes defined as hemoglobin A1c (HbA1c) >7.5%.
* Current medical history of drug or alcohol abuse within 12 months prior to screening.
* History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions, or severe allergic responses.
* Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.
* Subject has planned cardiac surgery, PCI or carotid stenting, or major non-cardiac surgery during the course of the study period or for 14 days after the last treatment.
* Use of any investigational drug in the 3 months prior to study drug administration.
* Use of insulin or any oral anti-diabetic (except metformin) in the 30 days prior to baseline measurements. Those subjects who are taking metformin may be included in the study if they are on a stable dose for at least 4 weeks and have a HbA1c <7.5%.
* Any contraindications for corticosteroid infusions (for example, but not limited current infections or vaccinations)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
18Fludeoxyglucose Positron emission computed tomography scan (18FDG PET-CT scan) | Day 8-13

CONTACTS AND LOCATIONS:
Overall Officials: Erik S Stroes, MD PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands